CLINICAL TRIAL: NCT04295382
Title: An Open-Label, Study of the Feasibility and the Usability of a Software Application to Deliver Targeted Interactive Exercises, in Addition to Treatment as Usual, to Patients Recently Hospitalized for Suicidal Ideation or Suicide Attempts
Brief Title: Feasibility Study of a Software Application for Patients Hospitalized After Suicidal Ideation or Suicide Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oui Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OUI-AVI-BT3
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Software Application (Experimental)
  Interventions: Device: Software Application

INTERVENTIONS:
Device: Software Application — A software application targeting suicidal ideation via interactive exercises.

SUMMARY:
The primary objective of this feasibility study is to assess the feasibility, and usability of a software application to deliver targeted interactive exercises to patients recently hospitalized for suicidal ideation or suicide attempts.

ELIGIBILITY:
Inclusion Criteria:

* English speaking male or female patients, 18-70 years
* Patients who have attempted suicide and voluntarily admitted themselves to an inpatient psychiatric unit or have clinically significant suicidal ideation and intent to harm themselves and are still on the inpatient psychiatric unit.
* Understand written and spoken English
* Own an iPhone with iOS 11 or higher, or Android with OS 8.1 or higher
* Willing and able to complete enrollment procedures
* Able to understand the nature of the study and provide written informed consent
* Able and willing to provide at least two verifiable contacts for emergency or tracking purposes.

Exclusion Criteria:

* Patients with active psychosis
* Patients who are acutely intoxicated at the time of enrollment
* Currently enrolled in other treatment studies for the symptoms and behaviors targeted
* Patients who are cognitively impaired
* Patients who, in the judgment of the investigator, would have an unfavorable risk/benefit (e.g. critically ill patients) profile with respect to the software application that delivers interactive exercises.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | 16 weeks
  The SUS is a valid and reliable, 10-item measure that effectively differentiates between usable and unusable systems. Sample items are "I think that I would like to use this app frequently" and "I felt very confident using the system." Responses are rated using a 5-point (strongly disagree to strongly agree) Likert scale. Scores range from 0 to 100, with a score of 68 being minimal indicator of usability.
User Feedback Interview Questions | 16 weeks
  Participants will answer the following questions. 1) What did you think about this experience? 2) Do you think you would use this app again if needed? Why (not)? 3) Do you think this app would be useful for helping you with your suicidal thoughts and preventing you from acting on them? Why (not)? Did you think functions were missing in the app? Which ones? 4) Is there anything else you think we should know to make this app better and more user-friendly?

SECONDARY OUTCOMES:
Suicidal ideation | 16 weeks
  The Beck Scale for Suicidal Ideation (BSS) is a 21-item self or clinician administered instrument used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide. Score range 0-42, with higher score indicating higher intensity.
Suicide attempts and other behaviors | 16 weeks
  This outcome will be assessed via the Columbia Suicide Severity Rating Scale (CSSRS), which was designed to classify suicide attempts, aborted suicide attempts, and other suicidal behaviors. Intensity of Ideation Subscale - includes 5 questions about the Frequency, Duration, Controllability, Deterrents, and Reasons for Ideation for the most severe level of ideation endorsed on the Severity subscale (i.e., highest endorsed from 1 to 5). The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk. Suicidal Behavior Lethality inquires about the level of actual medical damage or potential for it. Greater lethality or potential lethality of the behavior (endorsed on the Behavior subscale) indicates increased risk.
Diagnostic interview | 1 week
  The Mini International Neuropsychiatric Interview Neurocognitive (MINI) (40): this is a widely used, structured diagnostic interview that will be used to verify diagnosis at the screening visit.
Adverse events | 16 weeks
  The Systematic Assessment for Treatment Emergent Effects-Systematic Inquiry (SAFTEE-SI): This is a self-rated questionnaire assessing possible adverse events during the course of the trial. The purpose of the SAFTEE-SI is analytical and evaluates adverse events on a study level.
Depressive symptoms | 16 weeks
  The Patient Health Questionnaire (PHQ-9) is a 9-item self-report form to assess the severity of depressive symptoms that has been widely used in practice and research. This will be used throughout the study to assess severity of any depressive symptoms each participants is experiencing. The possible range is 0-27. Minimal depression (0-4). ≤ 4 The score suggests the patient may not need depression treatment. Mild depression (5-9). Moderate depression (10-14). 5 - 14 Physician uses clinical judgment about treatment, based on patient's duration of symptoms and functional impairment. Moderately severe depression (15-19). Severe depression (20-27). > 14 Warrants treatment for depression, using antidepressant, psychotherapy and/or a combination of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Wilkinson, M.D., Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No